CLINICAL TRIAL: NCT03336125
Title: Key Nutrients and Mental Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: Wisconsin Department of Health and Family Services (Other Government); Haukeland University Hospital (Other); National Institute of Nutrition and Seafood Research, Norway (Other Government)
Responsible Party: Principal Investigator, Anita Lill Hansen, Professor, University of Bergen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 983 974 724
Record Dates: First submitted 2017-10-26; First posted 2017-11-08 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Mental Health Impairment
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: Pre and post-test design
Who Masked: Participant
Masking Description: Double blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D group (Experimental): Intervention is vitamin D supplement
  Interventions: Dietary Supplement: Vitamin D
- Control group (Placebo Comparator): Placebo capsule contains olive oil
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D — Vitamin D (40µg/day) will be compared with placebo
  Arms: Vitamin D group
Dietary Supplement: Placebo — 120 mg olive oil
  Arms: Control group

SUMMARY:
The purpose of the project is to investigate whether an intervention program with vitamin D supplementation is able to improve the biology of stress resilience as well as subjective well-being in individuals with antisocial behavior problems (forensic inpatients).

DETAILED DESCRIPTION:
This is a randomized control trial looking at the effects of vitamin D supplements on mental health in a group of forensic inpatients. More specific the effects of vitamin D will be investigated in relation to underlying biological mechanisms associated with resilience (e.g., serotonin, cortisol, heart rate variability and executive functioning), but also subjective well-being such as sleep quality, anxiety, depression, self-reported resilience and physical activity. About 100 participants will be randomized to an intervention group (vitamin D) or a control group (placebo). The intervention will last for 3-4 months. Pre-test will start in October/November 2017 and post-test in April/May 2018.

ELIGIBILITY:
Inclusion Criteria:

* Patients with intelligence quotient > 70 will be invited.

Exclusion Criteria:

* Patients with intelligence quotient <70 will be excluded.
* Patients already taking vitamin D.
* Patients with psychotic disorders.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2018-05-22 (Actual); Study Completion 2018-05-22 (Actual)

PRIMARY OUTCOMES:
Change in vitamin D level in blood from pre-test (baseline) to post-test (after 4 months) | Time for blood sample: about 10-15 minutes (at both pre and post test)
  Measured from blood sample
Change in serotonin from pre-test (baseline) to post-test (after 4 months) | Time for blood sample: about 10-15 minutes (at both pre and post test)
  Measured form blood sample
Change in total cholesterol from pre-test (baseline) to post-test (after 4 months) | Time for blood sample: about 10-15 minutes (at both pre and post test)
  Measured from blood sample
Change in lipoproteins from pre-test (baseline) to post-test (after 4 months) | Time for blood sample: about 10-15 minutes (at both pre and post test)
  Measured from blood sample
Change in triglycerides from pre-test (baseline) to post-test (after 4 months) | Time for blood sample: about 10-15 minutes (at both pre and post-test)
  Measured from blood sample
Change in cortisol from pre-test (baseline) to post-test (after 4 months) | 7 samples over 24 hours (at both pre and post-test)
  Saliva
Change in performance on working memory tasks (N-back) from pre-test (baseline) to post-test (after 4 months) | About 8-10 minutes (at both pre and post-test)
  Computerized cognitive task
Change in performance on Tower of Hanoi Task from pre-test (baseline) to post-test (after 4 months) | About 10-15 minutes (at bot pre and post-test)
  Computerized cognitive task
Change in performance on Tower of London Task from pre-test (baseline) to post-test (after 4 months) | About 10-15 minutes (at both pre and post test)
  Computerized cognitive task
Change in performance on Iowa Gambling Task from pre-test (baseline) to post-test (after 4 months) | About 15-20 minutes (at both pre and post test)
  Computerized cognitive task
Change in heart rate variability from pre-test (baseline) to post-test (after 4 months) | 5 minutes of baseline, during the cognitive testing (up to 60 minutes) and 5 minutes of recovery (at both pre and post test)

SECONDARY OUTCOMES:
Change in sleep from pre-test (baseline) to post-test (after 4 months) | One week before intervention and one week after intervention (i.e., pre and post-test)
  Measured by Ambulatory Monitoring System together with a sleep log
Change on Epworth Sleepiness Scale from pre-test (baseline) to post-test (after 4 months) | About 5-10 minutes (at both pre and post-test)
Houston Non-Exercise Questionnaire | The physical activity log will be filled out weekly over the course of the study period (i.e., 24 -28 weeks) and estimated time per week is 10 minutes.
  The log consists of weekly recording of various activity levels.
Change in self-reported state and trait anxiety (STAI questionnaire) from pre-test (baseline) to post-test (after 4 months) | About 10 minutes (at both pre and post-test)
Change in self-reported resilience (Connor-Davidson Resilience Scale 25) from pre-test (baseline) to post-test (after 4 months) | About 5 minutes (at both pre and post-test)
Change in post-traumatic stress symptoms (Impact of event scale -Revised) from pre-test (baseline) to post-test (after 4 months) | About 5-10 minutes (at both pre and post-test)
Change in self-reported depression (Beck Depression Inventory) from pre-test (baseline) to post-test (after 4 months) | About 5-10 minutes (at both pre and post-test)

OTHER OUTCOMES:
Childhood Trauma Questionnaire | About 10 minutes (only at pre-test)
Iodine (test 1) | About 2-3 minutes
  Urin
Iodine (test 2) | About 2-3 minutes
  Urin

CONTACTS AND LOCATIONS:
Locations (1):
- Sand Ridge Secure Treatment Center, Mauston, Wisconsin, United States